CLINICAL TRIAL: NCT05905978
Title: Effectiveness and Safety of Donors Predisposed by Corneal Collagen Cross-linking in Deep Lamellar Keratoplasty for Treating the Patients With Keratoconus，A Randomized Controlled Trial.
Brief Title: Donors Predisposed by Corneal Collagen Cross-linking in Deep Lamellar Keratoplasty for the Patients With Keratoconus
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Zhongshan Ophthalmic Center, Sun Yat-sen University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2020KYPJ163
Record Dates: First submitted 2023-06-02; First posted 2023-06-15 (Actual); Last update posted 2023-06-15 (Actual); Status verified 2023-05

CONDITIONS: Keratoconus
Keywords: Corneal collagen cross-linking; Deep lamellar keratoplasty; Keratoconus
MeSH Terms: conditions — Keratoconus

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CXL graft group (Experimental): Corneal donors predisposed by CXL were used and the conventional DALK procedure was conducted in patients
  Interventions: Procedure: Corneal donors predisposed by CXL
- Conventional graft group (Active Comparator): Corneal donors stored in corneal storage media were used and the conventional DALK procedure was conducted in patients
  Interventions: Procedure: Corneal donors stored in corneal storage media

INTERVENTIONS:
Procedure: Corneal donors predisposed by CXL — Corneal donors predisposed by CXL and DALK procedure was conducted in patients
  Arms: CXL graft group
Procedure: Corneal donors stored in corneal storage media — Corneal donors stored in corneal storage media and DALK procedure was conducted in patients
  Arms: Conventional graft group

SUMMARY:
The Study was designed as a randomized controlled study with the following objectives:

To investigate whether use of donors predisposed by corneal collagen cross-linking (CXL) reduced myopic refractive errors for keratoconic eyes after Deep anterior lamellar keratoplasty (DALK).

Overall 70 patients are planned to recruit., the patients were assigned to CXL graft group, in which corneal donors predisposed by CXL were used, or the conventional graft group, in which corneal donors stored in corneal storage media were used. The patients will be followed-up for 24 months.

DETAILED DESCRIPTION:
Keratoconus is a progressive ecstatic corneal disease characterized by forward bulging of the cornea, thinning of the corneal stroma, and irregular astigmatism. Corneal transplantation is necessary for patients with advanced keratoconus when spectacles and contact lens are inadequate for visual correction. Deep anterior lamellar keratoplasty is a conventional procedure for the treatment of keratoconus. However, DALK itself frequently causes abnormality of refraction, such as high degrees of astigmatism owing to irregular corneal surface for keratoconic eyes. Possible mechanisms of this progressive astigmatism include the recurrence of keratoconus in the grafts, progressive corneal thinning of the host cornea, or progressive misalignment of the graft- host interface over time, which prevents the achievement of satisfactory vision.

Corneal collagen cross-linking is believed to have the ability to halt or decrease the progression of keratoconus. CXL treats keratoconus by strengthening corneal stromal collagen bonds with riboflavin activated by ultraviolet A (UVA), and is now a first-line treatment for progressive keratoconus. In this randomized controlled trial, we performed CXL on corneal donor tissues with the aim of achieving corneal stromal stiffening, thereafter DALK was conducted for the patients with advanced keratoconus using the tissues predisposed by CXL. The goal of this study is evaluating whether the strengthening grafts could reduce postoperative myopic refractive errors or arrest the progression of keratoconus for the patients with DALK.

ELIGIBILITY:
Inclusion Criteria:

* 1.The best corrected visual quality of frame glasses is less than 0.3，2.The best corrected visual quality of rigid gas permeable contact lens (RGPCL) is less than 0.5/ RGPCL intolerance，3.The anterior corneal surface curvature >55D，4.The thinnest corneal thickness is less than 400 μm. One of the above four items is met
* Patients must be willing and able to return for scheduled follow-up examinations for 36 months after surgery
* Ages：over 18 Years

Exclusion Criteria:

* History of intraocular surgery
* Severe dry eye
* Severe eyelid and conjunctival scar
* Loss of vision in contralateral eye
* Pregnant and lactating women

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2023-06 (Estimated); Primary Completion 2026-07 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Simulated keratometry | up to 36 months
  Simulated keratometry measured by topography

SECONDARY OUTCOMES:
Uncorrected distance visual acuity（UDVA） | 36 months
  UDVA (by using Snellen acuity charts) before surgery, at 1 week, 1, 3, 6, 9, 12, 15, 18, 21, 24, 30 and 36 months after surgery
Corrected distance visual acuity （CDVA） | 36 months
  CDVA (by using Snellen acuity charts) before surgery, at 1 week, 1, 3, 6, 9, 12, 15, 18, 21, 24, 30 and 36 months after surgery
Spherical equivalent (SE) | 36 months
  SE will be detected by combined optometry and phoroptor refractometer before surgery, at 1 week, 1, 3, 6, 9, 12, 15, 18, 21, 24, 30 and 36 months after surgery
Manifest cylinder | 36 months
  Manifest cylinder will be detected by topography before surgery, at 1 week, 1, 3, 6, 9, 12, 15, 18, 21, 24, 30 and 36 months after surgery
Corneal thickness | 36 months
  Corneal thickness of the thinnest area will be detected by Optical Coherence tomography before surgery, at 1 week, 1, 3, 6, 9, 12, 15, 18, 21, 24, 30 and 36 months after surgery
Corneal endothelium cells | 36 months
  Corneal endothelium cells will be detected by confocal microscopy before surgery, at 1 week, 1, 3, 6, 9, 12, 15, 18, 21, 24 ,30 and 36 months after surgery
Intraocular pressure | 36 months
  Intraocular pressure was measured by non-contact tonometer before surgery, at 1 week, 1, 3, 6, 9, 12, 15, 18, 21, 24,30 and 36 months after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongshan Ophthalmic Center, Sun Yat-Sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No